CLINICAL TRIAL: NCT05051371
Title: Incidence of Postoperative Residual Curarization in Elderly Patients in the Post-anesthesia Care Unit, and Attitude and Awareness Questionnaire of Anesthesiologists
Brief Title: Postoperative Residual Curarization in Elderly Patients in Post-anesthesia Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, aysun postaci, Ass. Prof. Dr. Nadide Aysun Postaci, Ankara City Hospital Bilkent
Other Study IDs: E1-21-1912
Record Dates: First submitted 2021-08-02; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Residual Curarization; Geriatrics
Keywords: Postoperative residual curarization; Geriatrics; Train of four
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Train of four monitoring — Train of four monitoring in postoperative care unit

SUMMARY:
In this study, we aimed to determine the knowledge levels and approaches of anesthesiologists working in our clinic about postoperative residual curarization(PORC) in elderly patients with a questionnaire. In addition, we aimed to determine the incidence of PORC and factors associated with PORC in the recovery unit in elderly patients over 65 years of age who underwent surgery under general anesthesia using muscle relaxants with a prospective observational study.

DETAILED DESCRIPTION:
Postoperative residual curarization (PORC) after general anesthesia is an important complication that can cause adverse patient outcomes, including symptoms of airway obstruction, hypoxia, respiratory distress, muscle weakness, and dyspnea in the early and late stages.

Anticholinesterase agents are commonly used to reverse neuromuscular blockade. Even with the use of anticholinesterase, severe PORC can be seen. The use of anticholinesterases in elderly patients is controversial due to the high side-effect profile.

Sugammadex, which has been widely used with its approval by the United States Food and Drug Administration in 2015, is a reverse agent that acts through a different mechanism than traditional anticholinesterase agents (it is a cyclodextrin molecule that encapsulates steroid neuromuscular blockers). Compared to neostigmine, sugammadex reverses neuromuscular blockade faster and more reliably.

In this study, we aimed to determine the knowledge levels and approaches of anesthesiologists working in our clinic about postoperative residual curarization(PORC) in elderly patients with a questionnaire. In addition, we aimed to determine the incidence of PORC and factors associated with PORC in the recovery unit in elderly patients over 65 years of age who underwent surgery under general anesthesia using muscle relaxants with a prospective observational study.

The first phase of the study is a prospective observational study. Elderly patients (>65) who are scheduled to undergo elective surgery under general anesthesia and require intubation using muscle relaxants will be screened for PORC using Train of four monitor in the recovery unit.

In the second phase of the study, an online questionnaire with 15 questions will determine the knowledge and attitudes of anesthesiologists working in our clinic on the use of muscle relaxants and reversing agents in elderly patients, the use of neuromuscular monitoring and PORC.

ELIGIBILITY:
Inclusion Criteria:

* age >65
* general anesthesia using non-depolarizing neuromuscular blocker

Exclusion Criteria:

* Patients with an ASA score greater than 3
* Those with contraindications to anesthetic drugs
* Those with neuromuscular, neurological and psychiatric diseases
* Patients in whom TOF monitoring is not possible in the ulnar nerve region
* Patients with advanced renal failure
* Patients with advanced hepatic insufficiency
* Those with decompensated heart failure
* Patients with BMI<18 and BMI>30
* Patients with uncontrolled hypertension, uncontrolled diabetes, pheochromocytoma, thyroid dysfunction
* Those who are incapable of reading and signing the consent form
* Patients who do not want to sign the consent form
* Patients deemed unsuitable by the investigator
* Those with chronic opioid use

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Electively operated elderly patients >65 years old under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative residual curarization | through study completion( anticipated 5 months)
  The incidence of elderly patients that Train of Four(TOF) rate <0.9 in the postoperative care unit

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Postaci, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided